CLINICAL TRIAL: NCT03151681
Title: Treating Adjustment Disorders Stemming From Romantic Betrayals: An Open-label Trial of Impairing Memory Reconsolidation Using Propranolol
Brief Title: The Trauma of Betrayal: Treating Adjustment Disorder With Reconsolidation Blockade Under Propranolol
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Alain Brunet, Ph.D., Primary Investigator and Full Professor, Department of Psychiatry, McGill University., Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRPL-006
Record Dates: First submitted 2017-04-29; First posted 2017-05-12 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Adjustment Disorders; Posttraumatic Stress Disorder; Trauma and Stressor Related Disorders
Keywords: Reconsolidation; Propranolol; Infidelity; Attachment injury; Romantic relationships
MeSH Terms: conditions — Adjustment Disorders; Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders | interventions — Propranolol

STUDY DESIGN:
Intervention Model Description: Experiment 1: Repeated measures open-label clinical trial with time-series analysis.
  Experiment 2: Randomized clinical trial (mismatch vs. no mismatch) with within-group wait-list.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization to 'mismatch group' or 'no-mismatch group' will be done prior to the first treatment session by a third party unrelated to the study, and blind to participant outcome. Participants will also be blind to which group they are randomized to. The randomization scheme will use the permuted-block method with a block size of four, stratified by gender (male and female) and event type (infidelity and other), and a group allocation probability of 50% (Fleiss, 1986).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propranolol pill + mismatch memory reactivation (Experimental): Prediction-error will be incorporated into each treatment sessions.
  Interventions: Drug: Propranolol Pill
- Propranolol pill + standard memory reactivation (Experimental)
  Interventions: Drug: Propranolol Pill
- Waitlist (No Intervention)

INTERVENTIONS:
Drug: Propranolol Pill — 1mg/kg of propranolol 60 minutes prior to memory reactivation
  Other Names: Inderal
  Arms: Propranolol pill + mismatch memory reactivation; Propranolol pill + standard memory reactivation

SUMMARY:
Attachment injuries are events occurring within couple relationships that involve betrayal or abandonment by a significant other during times of need (e.g., infidelity). They can be understood as relationship traumas, which can lead to debilitating symptoms consistent with posttraumatic stress disorder (PTSD), depression, and generalized anxiety for the injured partner. Research has demonstrated that the presence of an attachment injury represents a barrier to empirically effective couple's therapy. However, disrupting memory reconsolidation with the beta-blocker propranolol has been shown to alleviate PTSD symptoms by attenuating the salience of the emotional trauma memory, representing an interesting avenue for the treatment of adjustment disorders stemming from attachment injuries. Moreover, evidence suggests that a certain degree of mismatch, or an error between what is expected/predicted to occur and what actually occurs, must be present in order for a memory to destabilize and enter the reconsolidation phase following retrieval. Here, the investigators aim to extend the conditions under which reconsolidation therapy with propranolol can be used in a clinical setting, as well as assess whether incorporating mismatch enhances treatment effects. The investigators hypothesize that, compared to a wait-list control, 4-6 sessions of memory reactivation under propranolol will significantly reduce trauma-related and general anxio-depressive symptoms, associated with an attachment injury. Moreover, the investigators hypothesize that participants randomized to the mismatch group will improve significantly more than the standard treatment group on all variables of interest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an adjustment disorder or chronic adjustment disorder, as defined by the Diagnostic and Statistical Manual for Mental Disorders, as a result of an attachment injury, defined as an event involving the perceived betrayal, violation of trust, or abandonment by a significant other.
* Currently experiencing clinically important psychological distress as a result of the event, as defined by a score of at least 22 on the IES-R, and a score of at least "moderately ill" on the Clinical Global Impressions - Severity of Illness Scale.
* Must have been in the romantic relationship for at least 6 months prior to the event.
* Must not take psychotropic medication.
* Fluency in English or French

Exclusion Criteria:

* Systolic blood pressure <100 mm Hg;
* Cardiac rhythm below 55 beats per minute;
* A medical condition that contraindicates the administration of propranolol, e.g., Asthma, chronic obstructive pulmonary disease, cardiac insufficiency, cardiac choc, Second- or third-degree atrioventricular block, diabetes, spastic angina, auricular sinus illness, bradycardia, Raynaud's disease, severe peripheral vascular disease, untreated Pheochromocytoma, arterial hypotension, previous anaphylactic allergic shock;
* Previous adverse reaction to, or non-compliance with, beta-blocker;
* Current use of a substance that may involve potentially dangerous interactions with propranolol, including P450 2D6 inhibitors.
* Women who are pregnant or breast feeding;
* Individuals currently participating in any other form of psychotherapy (other than strictly supportive).
* History of substance dependence disorder, bipolar disorder, or psychotic disorder;
* Participants judged (based on history, mental status exam, clinical impression, or the Suicidal Behaviors Questionnaire as being at significant risk of suicidal behavior.
* Participation in another drug trial within 30 days prior to the screening visit
* Presence of any clinical condition that might interfere with the interpretation of the efficacy and safety results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Within-group difference: Wait-list vs. Treatment; Between-group difference: Mismatch vs. No Mismatch on Impact of Events Scale-Revised | Administered at baseline (Week 0), Post-Wait-list (Week 4), at each subsequent weekly visit, at the one-week post-treatment follow-up, and at the three-month follow up.
  Severity of Trauma and Stressor-related symptoms

SECONDARY OUTCOMES:
Within-group difference: Wait-list vs. Treatment; Between-group difference: Mismatch vs. No Mismatch on Hopkins Symptom Checklist-25 | Administered at baseline (Week 0), Post-Wait-list (Week 4), at each subsequent weekly visit, at the one-week post-treatment follow-up, and at the three-month follow up.
  General Psychological Distress (Depression and Anxiety)
Within-group difference: Wait-list vs. Treatment; Between-group difference: Mismatch vs. No Mismatch on World Health Organization - Quality of Life BREF | Administered at baseline (Week 0), Post-Wait-list (Week 4), at the one-week post-treatment follow-up, and at the three-month follow up.
  Perceived Quality of Life in 4 Domains, Psychological, Physical, Environmental, Social

CONTACTS AND LOCATIONS:
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lonergan M, Saumier D, Pigeon S, Etienne PE, Brunet A. Treatment of adjustment disorder stemming from romantic betrayal using memory reactivation under propranolol: A open-label interrupted time series trial. J Affect Disord. 2022 Nov 15;317:98-106. doi: 10.1016/j.jad.2022.08.082. Epub 2022 Aug 27. PMID 36031005